CLINICAL TRIAL: NCT02988141
Title: A Prospective Multi-center Study to Investigate the EGFR-TKI Resistance Profile in Chinese Patients With Advanced EGFRm+ NSCLC
Brief Title: EGFR-TKI Resistance Profile in Chinese Patients With Advanced EGFRm+ NSCLC
Acronym: PRECENT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jianxing He (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Jianxing He, Principle Investigator, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: CCTC1601
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — ctDNA in blood and tissues
Oversight: Data Monitoring Committee: No

SUMMARY:
A Prospective Multi-center Study to Investigate the EGFR-TKI Resistance Profile in Chinese Patients with Advanced EGFRm+ NSCLC

DETAILED DESCRIPTION:
Patients with EGFR mutation and presented secondary resistance to prior first-generation EGFR-TKI should have received biopsy of at least on progressed lesions and are able to provide tissues for pathological examination and NGS testing.All enrolled patients will be followed up to clinical outcome (treatments, tumor response, survival, etc).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Male or female patients aged 18 years and older.
* Histological confirmation of stage IIIB/IV NSCLC.
* Documented EGFR mutation positive .
* WHO Performance Status 0, 1 or 2

Exclusion Criteria:

* Any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study.
* Previous (within 6 months) or current treatment with AZD9291.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EGFR mutation positive patients with paired tissue and blood samples
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
The biomarker profile of EGFR-TKI resistance | Baseline

SECONDARY OUTCOMES:
The concordance, sensitivity and specificity in paired blood and tissue samples | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jian Xing HE, MD, Principal Investigator — China

IPD SHARING:
Plan to Share IPD: No